CLINICAL TRIAL: NCT03548064
Title: A Phase 1 Double-Blinded, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety and Immunogenicity of Double Mutant Heat-Labile Toxin LTR192G/L211A (dmLT) From Enterotoxigenic Escherichia Coli (ETEC) by Oral, Sublingual, or Intradermal Vaccination in Adults Residing in an Endemic Area
Brief Title: A Double-Blind Placebo-Control Dose Escalating Study to Evaluate the Safety and Immunogenicity of dmLT by Oral, Sublingual and Intradermal Vaccination in Adults Residing in an Endemic Area
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID 19 cases at the site
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 14-0031
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Results first posted 2022-01-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2017-12-14

CONDITIONS: Gastroenteritis Escherichia Coli; Immunisation
Keywords: dmLT; E. coli; Enterotoxigenic Escherichia coli (ETEC); LTR192G/L211A
MeSH Terms: conditions — Escherichia coli Infections | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Regimen A (Experimental): 5 µg of dmLT oral on days 1, 15, 29, n=12; placebo oral on days 1, 15, 29, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen B (Experimental): 25 µg of dmLT oral on days 1, 15, 29, n=12; placebo oral on days 1, 15, 29, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen C (Experimental): 5 µg of dmLT sublingual on days 1, 15, 29, n=12; placebo sublingual on days 1, 15, 29, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen D (Experimental): 25 µg of dmLT sublingual on days 1, 15, 29, n=12; placebo sublingual on days 1, 15, 29, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen E (Experimental): 0.3 µg of dmLT intradermal on days 1, 22, 43, n=12; placebo intradermal on days 1, 22, 43, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen F (Experimental): 1.0 µg of dmLT intradermal on days 1, 22, 43, n=12; placebo intradermal on days 1, 22, 43, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen G (Experimental): 50 µg of dmLT oral on days 1, 15, 29, n=12; placebo oral on days 1, 15, 29, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen H (Experimental): 50 µg of dmLT sublingual on days 1, 15, 29, n=12; placebo sublingual on days 1, 15, 29, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine
- Regimen I (Experimental): 2.0 µg of dmLT intradermal on days 1, 22, 43, n=12; placebo intradermal on days 1, 22, 43, n=3
  Interventions: Other: Placebo; Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine

INTERVENTIONS:
Other: Placebo — Placebo
  Arms: Regimen A; Regimen B; Regimen G
Other: Placebo — Placebo
  Arms: Regimen C; Regimen D; Regimen H
Other: Placebo — Placebo
  Arms: Regimen E; Regimen F; Regimen I
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
  Arms: Regimen A; Regimen B; Regimen G
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
  Arms: Regimen C; Regimen D; Regimen H
Biological: Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) Oral enterotoxigenic Escherichia coli (ETEC) Vaccine — LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
  Arms: Regimen E; Regimen F; Regimen I

SUMMARY:
This is a trial to evaluate the safety and immunogenicity of double mutant heat-labile toxin LTR192G/L211A (dmLT) from Enterotoxigenic Escherichia coli (ETEC) by oral, sublingual, or intradermal vaccination in approximately 135 healthy adult volunteers, age 18-45 years. Study duration is approximately 2.5 years, with each participant duration for up to 9 months depending on the route of dmLT administered. There is no specific hypothesis being tested in this study. The primary objective of this study is to assess the reactogenicity, safety, and tolerability of dmLT when administered in three sequential doses, over a range of dosages by oral, sublingual, or intradermal routes.

DETAILED DESCRIPTION:
This is a Phase 1 double-blinded, placebo-controlled, dose-escalation trial to evaluate the safety and immunogenicity of double mutant heat-labile toxin LTR192G/L211A (dmLT) from Enterotoxigenic Escherichia coli (ETEC) by oral, sublingual, or intradermal vaccination in approximately 135 healthy adult volunteers, age 18-45 years, who meet all the eligibility criteria and reside in Bangladesh. Study duration is approximately 2.5 years, with each participant duration for up to 9 months depending on the route of dmLT administered. The study population will be recruited from Mirpur, a community of Dhaka, Bangladesh, known as having a high rate of diarrheal, respiratory, and enteric disease. This clinical trial is designed to assess the safety, reactogenicity, tolerability, and immunogenicity of a range of dosages of dmLT administered by three different routes: oral, sublingual, or intradermal. The oral and sublingual routes of administration will evaluate dosages of 5, 25, and 50 micrograms of dmLT; the intradermal route of administration will evaluate dosages of 0.3, 1.0, and 2.0 micrograms of dmLT. Participants will receive a total of three sequential doses of dmLT; the oral and sublingual routes will be at days 1, 15, and 29 and the intradermal route will be at days 1, 22, and 43. There is no specific hypothesis being tested in this study. The primary objective of this study is to assess the reactogenicity, safety, and tolerability of dmLT when administered in three sequential doses, over a range of dosages by oral, sublingual, or intradermal routes. The secondary objectives of this study are: 1) to assess the long-term safety, from first vaccination through 6 months following the last dose of vaccine, 2) to evaluate the serum anti-dmLT IgG and IgA response, 3) to evaluate the IgG and IgA anti-dmLT Antibody Secreting Cell (ASC) response, 4) to evaluate the IgG and IgA anti-dmLT Antibodies in Lymphocyte Supernatant (ALS) response, 5) to evaluate the total fecal IgA and fecal anti-dmLT IgA response, and 6) to evaluate the total salivary IgA and the saliva-derived anti-dmLT IgA response.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18-45 years old, inclusive.
2. Provides written informed consent before initiation of any study procedures.
3. Healthy as judged by the site investigators and determined by medical history, medication history, and physical examination.
4. Capable of understanding, consenting, and complying with all the study visits and procedures.
5. Body Mass Index of no less than 18.5.
6. Agrees not to participate in another clinical trial during the study period.
7. Agrees to complete all study visits and procedures.
8. Agrees not to donate blood to a blood bank for 12 months after receiving the last vaccine.

Exclusion Criteria:

1. Women who are pregnant or lactating or have a positive urine pregnancy test at screening or on the day of vaccinations.

   Note: all women presenting for screening will have urine pregnancy testing. "Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control from screening and through 28 days post last dose of vaccine. Abstinence is also acceptable."
2. Presence or history of a chronic medical condition* that would, in the opinion of the investigator, render vaccination unsafe or interfere with the evaluation of the vaccine.

   *Note: this may include, but is not limited to: significant renal disease, unstable or progressive neurological disorders, diabetes, heart disease, asthma, lung disease, liver disease, organ transplant recipients and cancer.
3. Presence of a significant dermatologic condition*, or tattoo(s), scarring or significant skin damage at the vaccination site that would impede evaluation of local reactogenicity.

   *Note: this may include severe eczema, psoriasis or history of keloid formation. Participants with history of squamous cell or basal cell skin cancer that has been surgically excised and considered cured may be enrolled in the study if the skin cancer site is healed and is not at proposed vaccine administration site.
4. Any developmental abnormality of the palate.
5. Participants diagnosed with autoimmune disorders, chronic inflammatory disorders or neurological disorders with a potential autoimmune correlation.
6. Use of long-term (> / = 2 weeks) oral steroids, intranasal or topical prednisone (or equivalent), parenteral steroids, or high-dose inhaled steroids (> 800 microgram/day of beclomethasone dipropionate or equivalent) within the preceding 6 months.
7. Has major psychiatric illness* during last 12 months that in the investigator's opinion would preclude participation.

   *Note: Participants taking antipsychotic or antimanic drugs should not be enrolled. These include: aripiprazole, clozapine, ziprasidone, haloperidol, molindone, lamotrigine, gabapentin, topiramate, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate, or lithium citrate. Participants taking a single antidepressant drug and are stable without de-compensating symptoms in the preceding 3 months can be enrolled in the study.
8. Use of prescription or over-the-counter (OTC) anti-inflammatory medications* 48 hours prior to receiving the investigational product.

   *Note: This includes naproxen, aspirin, ibuprofen, and other non-steroidal anti-inflammatory drugs.
9. Gastrointestinal symptoms* in the past 24 hours or abdominal pain lasting for more than 2 weeks in the past 6 months.

   *Note: this may include, but is not limited to: abdominal pain or cramps, loss of appetite, nausea, general ill-feeling or vomiting.
10. Moderate or severe diarrheal illness* during the 6 weeks prior to enrollment.

    *Note: Moderate or severe diarrheal illness is defined by the passage of > / = 4 unformed or loose stools (mix of liquid and solid components) in a 24 hour period
11. History of chronic gastrointestinal illness*.

    *Note: this includes severe dyspepsia or gastroesophageal reflux disease, constipation, irritable bowel syndrome (IBS), hemorrhoids, diverticular disease, colitis, colon polyps, colon cancer, and inflammatory bowel disease. Mild or moderate heartburn or epigastric pain occurring no more than three times per week is permitted.
12. Regular use (weekly or more often) of laxatives, anti-diarrheal, anti-constipation, or antacid therapy.
13. History of major gastrointestinal surgery, excluding uncomplicated appendectomy or cholecystectomy.
14. History of systemic antimicrobial treatment (i.e., topical treatments are not an exclusion) during the week prior to any administration of dmLT.
15. Acute febrile illness (body temperature > / = 38 degrees Celsius) during the week prior to enrollment.
16. Abnormal screening laboratories. Note: screening labs include white blood cell count (WBC), absolute neutrophil count (ANC), hemoglobin (Hg), platelet count, serum creatinine, serum albumin, alanine aminotransferase (ALT, also known as SGPT), and serologic testing for Hepatitis B virus surface antigen (HBsAg) and Hepatitis C virus (HCV) antibody. Abnormal vital signs.
17. Isolation of specific bacteria* from screening stool cultures.

    *Note: bacteria include ETEC, Vibrio cholerae, and Shigella spp. Salmonella and Campylobacter will not be evaluated as part this criterion.
18. Received an inactivated licensed vaccine within 2 weeks of enrollment or live licensed vaccine within 4 weeks of enrollment.
19. Received a cholera (licensed or experimental) vaccine, E. coli vaccine, or Shigella vaccine in the last 3 years.
20. History of receiving immune globulin or other blood product within the 3 months before enrollment in this study.
21. Currently enrolled in another study, involving an experimental agent. Participants involved in observational studies or surveys remain eligible.
22. Any condition that would, in the opinion of the Site Investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.
23. Known allergies to study compound or components of the study vaccine.
24. Donating blood in the 8 weeks prior to study entry.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States
- International Center for Diarrheal Disease Research Bangladesh - Infectious Diseases Division - Mucosal Immunology and Vaccinology Unit, Dhaka, Bangladesh

REFERENCES:
- [Derived] Bhuiyan TR, Khanam F, Basher SR, Dash P, Chowdhury MI, Haque S, Harun NB, Akter A, Karmakar PC, Hakim A, Amin S, Kamruzzaman M, Parvin N, Ahmed T, Butts J, Pasetti MF, Wahid R, Sztein MB, Maier N, White JA, Tomashek KM, Bourgeois AL, Baqar S, Kotloff KL, Qadri F, Chen WH. Safety and immunogenicity of a recombinant double-mutant heat-labile toxin derived from enterotoxigenic Escherichia coli in healthy Bangladeshi adults delivered by three different routes. Front Bacteriol. 2025;4:10.3389/fbrio.2025.1567791. doi: 10.3389/fbrio.2025.1567791. Epub 2025 Jul 15. PMID 41306922

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females between 18 and 45 years old, inclusively. They were recruited from the community at large around the clinic site. The enrollment period occurred between 10MAR2019 and 11FEB2020.
Groups:
- Oral 5 µg dmLT: 5 µg of dmLT administered orally on Days 1, 15, and 29.
  Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) enterotoxigenic Escherichia coli (ETEC) Vaccine: LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
- Oral 25 µg of dmLT: 25 µg of dmLT administered orally on Days 1, 15, and 29.
  Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) enterotoxigenic Escherichia coli (ETEC) Vaccine: LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
- Oral Placebo: Placebo administered orally on Days 1, 15, and 29.
  Placebo: Sodium bicarbonate buffer is a solution of 2 g sodium bicarbonate in 150 mL of sterile water for injection.
- Sublingual 5 µg of dmLT: 5 µg of dmLT administered sublingually on Days 1, 15, and 29.
  Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) enterotoxigenic Escherichia coli (ETEC) Vaccine: LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
- Sublingual 25 µg of dmLT: 25 µg of dmLT administered sublingually on Days 1, 15, and 29.
  Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) enterotoxigenic Escherichia coli (ETEC) Vaccine: LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
- Sublingual Placebo: Placebo administered sublingually on Days 1, 15, and 29.
  Placebo: 0.9% Sodium Chloride, USP (Normal Saline) is a sterile, nonpyrogenic, isotonic solution of sodium chloride 9 mg and may contain hydrochloric acid and/or sodium hydroixde for pH adjustment (pH 5.3, range 4.5 - 7.0).
- Intradermal 0.3 µg of dmLT: 0.3 µg of dmLT administered intradermally on Days 1, 22, and 43. Recombinant Double Mutant Heat-Labile Toxin LT(R192G/L211A) (dmLT) enterotoxigenic Escherichia coli (ETEC) Vaccine: LT(R192G/L211A), or dmLT is a derivative of wild-type enterotoxigenic Escherichia coli heat-labile enterotoxin that has been genetically modified by replacing the arginine at amino acid position 192 with glycine and the leucine at amino acid position 211 with alanine. These two amino acid substitutions take place in proteolytic cleavage sites which are critical for activation of the secreted toxin molecules.
- Intradermal Placebo: Placebo administered intradermally on Days 1, 22, and 43.
  Placebo: 0.9% Sodium Chloride, USP (Normal Saline) is a sterile, nonpyrogenic, isotonic solution of sodium chloride 9 mg and may contain hydrochloric acid and/or sodium hydroixde for pH adjustment (pH 5.3, range 4.5 - 7.0).
Period: Overall Study
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Started | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3
Completed | 12 | 12 | 6 | 11 | 0 | 3 | 12 | 3
Not Completed | 0 | 0 | 0 | 1 | 12 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Covid-19 Pandemic | 0 | 0 | 0 | 0 | 10 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo | Total
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (6.6) | 28.8 (7.0) | 25.5 (4.9) | 27.8 (7.1) | 28.8 (7.4) | 32.7 (5.9) | 31.0 (7.4) | 35.0 (3.6) | 29.6 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 5 | 8 | 2 | 6 | 2 | 38
  Male | 8 | 5 | 2 | 7 | 4 | 4 | 6 | 1 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3 | 75
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bangladesh | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3 | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in the Oral Arms With Solicited Local Reactogenicity Events Post Each Dose
Description: Solicited adverse events were collected post-vaccination and for 7 days after. Local events for the oral route include irritation of the oral cavity or tongue, diarrhea, nausea, vomiting, and abdominal discomfort.
Time Frame: Day 1 through Day 8 (post dose 1), Day 15 through Day 22 (post dose 2), Day 29 through Day 36 (post dose 3)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Oral 5 µg dmLT: 5 µg of dmLT administered orally on Days 1, 15, and 29.
- Oral 25 µg dmLT: 25 µg of dmLT administered orally on Days 1, 15, and 29.
- Oral Placebo: Placebo administered orally on Days 1, 15, and 29.
Arm/Group | Oral 5 µg dmLT | Oral 25 µg dmLT | Oral Placebo
Number analyzed (Participants) | 12 | 12 | 6
Participants
  Post Dose 1: Irritation of oral cavity or tongue | 0 | 0 | 0
  Post Dose 1: Diarrhea | 0 | 0 | 0
  Post Dose 1: Nausea | 0 | 0 | 0
  Post Dose 1: Vomiting | 0 | 0 | 0
  Post Dose 1: Abdominal discomfort | 0 | 0 | 0
  Post Dose 1: None | 12 | 12 | 6
  Post Dose 2: Irritation of oral cavity or tongue | 0 | 0 | 0
  Post Dose 2: Diarrhea | 0 | 0 | 0
  Post Dose 2: Nausea | 0 | 0 | 0
  Post Dose 2: Vomiting | 0 | 3 | 0
  Post Dose 2: Abdominal discomfort | 0 | 0 | 0
  Post Dose 2: None | 12 | 9 | 6
  Post Dose 3: number analyzed (Participants) | 11 | 12 | 6
  Post Dose 3: Irritation of oral cavity or tongue | 0 | 0 | 0
  Post Dose 3: Diarrhea | 0 | 0 | 0
  Post Dose 3: Nausea | 0 | 0 | 0
  Post Dose 3: Vomiting | 0 | 0 | 0
  Post Dose 3: Abdominal discomfort | 0 | 0 | 0
  Post Dose 3: None | 11 | 12 | 6

2. Primary Outcome: Number of Participants in the Sublingual Arms With Solicited Local Reactogenicity Events Post Each Dose
Description: Solicited adverse events were collected post-vaccination and for 7 days after. Local events for the sublingual route include irritation of the oral cavity or tongue, facial nerve disturbance, diarrhea, nausea, vomiting, or abdominal discomfort.
Time Frame: Day 1 through Day 8 (post dose 1), Day 15 through Day 22 (post dose 2), Day 29 through Day 36 (post dose 3)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Sublingual 5 µg of dmLT: 5 µg of dmLT administered sublingually on Days 1, 15, and 29.
- Sublingual 25 µg of dmLT: 25 µg of dmLT administered sublingually on Days 1, 15, and 29.
- Sublingual Placebo: Placebo administered sublingually on Days 1, 15, and 29.
Arm/Group | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo
Number analyzed (Participants) | 12 | 12 | 6
Participants
  Post Dose 1: Irritation of oral cavity or tongue | 0 | 0 | 0
  Post Dose 1: Facial nerve disturbance | 0 | 0 | 0
  Post Dose 1: Diarrhea | 0 | 0 | 0
  Post Dose 1: Nausea | 0 | 0 | 0
  Post Dose 1: Vomiting | 0 | 0 | 0
  Post Dose 1: Abdominal discomfort | 0 | 0 | 0
  Post Dose 1: None | 12 | 12 | 6
  Post Dose 2: number analyzed (Participants) | 12 | 10 | 6
  Post Dose 2: Irritation of oral cavity or tongue | 0 | 0 | 0
  Post Dose 2: Facial nerve disturbance | 0 | 0 | 0
  Post Dose 2: Diarrhea | 0 | 0 | 0
  Post Dose 2: Nausea | 0 | 0 | 0
  Post Dose 2: Vomiting | 0 | 0 | 0
  Post Dose 2: Abdominal discomfort | 0 | 0 | 0
  Post Dose 2: None | 12 | 10 | 6
  Post Dose 3: number analyzed (Participants) | 12 | 10 | 6
  Post Dose 3: Irritation of oral cavity or tongue | 0 | 0 | 0
  Post Dose 3: Facial nerve disturbance | 0 | 0 | 0
  Post Dose 3: Diarrhea | 0 | 0 | 0
  Post Dose 3: Nausea | 0 | 0 | 0
  Post Dose 3: Vomiting | 0 | 0 | 0
  Post Dose 3: Abdominal discomfort | 0 | 0 | 0
  Post Dose 3: None | 12 | 10 | 6

3. Primary Outcome: Number of Participants in the Intradermal Arms With Solicited Local Reactogenicity Events Post Each Dose
Description: Solicited adverse events were collected post-vaccination and for 7 days after. Local events for the intradermal route include injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, vesicles, or hardened mass.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 1 through Day 8 (post dose 1), Day 22 through Day 29 (post dose 2)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Intradermal 0.3 µg dmLT: 0.3 µg of dmLT administered intradermally on Days 1, 22, and 43.
- Intradermal Placebo: Placebo administered intradermally on Days 1, 22, and 43.
Arm/Group | Intradermal 0.3 µg dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 3
Participants
  Post Dose 1: Injection site pain | 0 | 0
  Post Dose 1: Injection site redness | 2 | 0
  Post Dose 1: Injection site swelling | 0 | 0
  Post Dose 1: Injection site bruising | 0 | 0
  Post Dose 1: Injection site pruritus | 0 | 0
  Post Dose 1: Injection site hypopigmentation | 0 | 0
  Post Dose 1: Injection site hyperpigmentation | 0 | 0
  Post Dose 1: Injection site induration | 1 | 0
  Post Dose 1: Injection site vesicles | 0 | 0
  Post Dose 1: Injection site mass | 0 | 0
  Post Dose 1: None | 9 | 3
  Post Dose 2: Injection site pain | 0 | 0
  Post Dose 2: Injection site redness | 0 | 0
  Post Dose 2: Injection site swelling | 0 | 0
  Post Dose 2: Injection site bruising | 0 | 0
  Post Dose 2: Injection site pruritus | 0 | 0
  Post Dose 2: Injection site hypopigmentation | 0 | 0
  Post Dose 2: Injection site hyperpigmentation | 0 | 0
  Post Dose 2: Injection site induration | 0 | 0
  Post Dose 2: Injection site vesicles | 0 | 0
  Post Dose 2: Injection site mass | 0 | 0
  Post Dose 2: None | 12 | 3

4. Primary Outcome: Number of Participants in the Oral and Sublingual Arms With Solicited Systemic Reactogenicity Events Post Each Dose
Description: Solicited adverse events were collected post-vaccination and for 7 days after. Systemic events for the oral and sublingual routes include fever, feverishness, fatigue, malaise, myalgia, or headache.
Time Frame: Day 1 through Day 8 (post dose 1), Day 15 through Day 22 (post dose 2), Day 29 through Day 36 (post dose 3)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Oral 25 µg of dmLT: 25 µg of dmLT administered orally on Days 1, 15, and 29.
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 6
Participants
  Post Dose 1 | 3 | 1 | 0 | 0 | 0 | 1
  Post Dose 2: number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6
  Post Dose 2 | 1 | 0 | 0 | 1 | 0 | 0
  Post Dose 3: number analyzed (Participants) | 11 | 12 | 6 | 12 | 10 | 6
  Post Dose 3 | 1 | 0 | 0 | 1 | 0 | 0

5. Primary Outcome: Number of Participants in the Intradermal Arms With Solicited Systemic Reactogenicity Events Post Each Dose
Description: Solicited adverse events were collected post-vaccination and for 7 days after. Systemic events for the intradermal route include fever, feverishness, fatigue, malaise, myalgia, headache, diarrhea, nausea, vomiting, or abdominal discomfort.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 1 through Day 8 (post dose 1), Day 22 through Day 29 (post dose 2)
Population: The Safety Analysis population includes all participants who received at least one study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Intradermal 0.3 µg dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 3
Participants
  Post Dose 1 | 0 | 0
  Post Dose 2 | 0 | 0

6. Primary Outcome: Number of Participants Who Withdrew From the Study
Description: Participants could voluntarily withdraw their consent for study participation for any reason at any time. Primary reason for withdrawal was recorded and early termination visits were attempted.
Time Frame: Day 1 through Day 209 (Day 223 for Intradermal cohorts)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Groups:
- Intradermal 0.3 µg of dmLT: 0.3 µg of dmLT administered intradermally on Days 1, 22, and 43.
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3
Participants | 0 | 0 | 0 | 1 | 12 | 3 | 0 | 0

7. Primary Outcome: Number of Participants Who Discontinued Study Vaccination
Description: Participants who received the first vaccination could choose to discontinue receipt of study vaccine for any reason and could choose to remain in the study (i.e., not withdraw from study). In addition, a participant could be discontinued from receipt of the second or third vaccination. Discontinuation from vaccination did not mean automatic withdrawal from the study, and participants were monitored for safety and immunogenicity if the participant consented.
Time Frame: Day 1 through Day 29 (Day 43 for Intradermal cohorts)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3
Participants | 1 | 0 | 0 | 0 | 2 | 0 | 12 | 3

8. Primary Outcome: Number of Vaccine-related Unsolicited Adverse Events From First Dose Through 28 Days After Last Dose
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment.
Time Frame: Day 1 through Day 57 (Day 71 for Intradermal cohorts)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3
Participants
  Mild (Grade 1) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Moderate (Grade 2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Vaccine-related Serious Adverse Events From Post Dose 1 Through 6 Months After Last Dose
Description: Serious Adverse Events (SAE) were defined as an adverse event which resulted in death, was life threatening, resulted in an inpatient hospitalization, prolongation of an existing hospitalization, led to persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or led to a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalizations were considered serious when, based upon appropriate medical judgment, they jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 209 (Day 223 for Intradermal cohorts)
Population: The Safety Analysis population includes all participants who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 12 | 6 | 12 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With a >= 4-fold Rise in dmLT-specific Serum IgA Titers Over Baseline Measured by ELISA
Description: Blood was collected for the IgA and IgG assay which was conducted with dmLT as the antigen. Each sample was tested per the laboratory's standard operating procedure. The percentage of participants with a >= 4-fold rise in dmLT-specific serum IgA and IgG titers over baseline was calculated for each study arm from the available results at any time post-first study vaccination.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 8 through Day 114
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Post-Dose 1 Day 7 (Day 8) | 0 [0 to 26.5] | 42 [15.2 to 72.3] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 70.8]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 8 [0.2 to 38.5] | 67 [34.9 to 90.1] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 75 [42.8 to 94.5] | 0 [0 to 70.8]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 0 [0 to 26.5] | 83 [51.6 to 97.9] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] | 83 [51.6 to 97.9] | 0 [0 to 70.8]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 17 [2.1 to 48.4] | 75 [42.8 to 94.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 0 [0 to 26.5] | 67 [34.9 to 90.1] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 28 (Day 57 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 11 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 28 (Day 57 oral/sublingual) | 0 [0 to 26.5] | 33 [9.9 to 65.1] | 0 [0 to 45.9] | 0 [0 to 28.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 85 (Day 114 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 11 | 0 | 3 | 0 | 0
  Post-Dose 3 Day 85 (Day 114 oral/sublingual) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 28.5] |  | 0 [0 to 70.8] |  |

11. Secondary Outcome: Percentage of Participants With a >= 4-fold Rise in dmLT-specific Serum IgG Titers Over Baseline Measured by ELISA
Description: Blood was collected for the IgG and IgA assay which was conducted with dmLT as the antigen. Each sample was tested per the laboratory's standard operating procedure. The percentage of participants with a >= 4-fold rise in dmLT-specific serum IgG and IgA titers over baseline was calculated for each study arm from the available results at any time post-first study vaccination.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 8 through Day 114
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Post-Dose 1 Day 7 (Day 8) | 8 [0.2 to 38.5] | 17 [2.1 to 48.4] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 70.8]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 17 [2.1 to 48.4] | 67 [34.9 to 90.1] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 67 [34.9 to 90.1] | 0 [0 to 70.8]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 25 [5.5 to 57.2] | 83 [51.6 to 97.9] | 0 [0 to 45.9] | 0 [0 to 26.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] | 75 [42.8 to 94.5] | 0 [0 to 70.8]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 25 [5.5 to 57.2] | 83 [51.6 to 97.9] | 0 [0 to 45.9] | 0 [0 to 26.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 25 [5.5 to 57.2] | 83 [51.6 to 97.9] | 0 [0 to 45.9] | 0 [0 to 26.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 28 (Day 57 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 11 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 28 (Day 57 oral/sublingual) | 33 [9.9 to 65.1] | 92 [61.5 to 99.8] | 0 [0 to 45.9] | 0 [0 to 28.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 85 (Day 114 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 11 | 0 | 3 | 0 | 0
  Post-Dose 3 Day 85 (Day 114 oral/sublingual) | 25 [5.5 to 57.2] | 50 [21.1 to 78.9] | 0 [0 to 45.9] | 0 [0 to 28.5] |  | 0 [0 to 70.8] |  |

12. Secondary Outcome: Percentage of Participants With >= 8 dmLT-specific IgA ASC / 10^6 PBMC as Measured by ELISpot
Description: PBMCs were collected for the IgA and IgG assay which was conducted with dmLT as the antigen. Each sample was tested per the laboratory's standard operating procedure. The percentage of participants with >= 8 dmLT-specific IgA and IgG ASC / 10^6 PBMC was calculated for each study arm from the available results at any time post-first study vaccination.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 1 through Day 36
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination blood sample for immunogenicity testing for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Pre-Dose 1 (Day 1): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 9 | 2
  Pre-Dose 1 (Day 1) | 0 [0 to 26.5] | 8 [0.2 to 38.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 0 [0 to 33.6] | 0 [0 to 84.2]
  Post-Dose 1 Day 7 (Day 8) | 0 [0 to 26.5] | 25 [5.5 to 57.2] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 17 [2.1 to 48.4] | 0 [0 to 70.8]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 70.8]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 0 [0 to 26.5] | 8 [0.2 to 38.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 42 [15.2 to 72.3] | 0 [0 to 70.8]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] |  |

13. Secondary Outcome: Percentage of Participants With >= 8 dmLT-specific IgG ASC / 10^6 PBMC as Measured by ELISpot
Description: as for outcome 12
Time Frame: Day 1 through Day 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Pre-Dose 1 (Day 1): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 9 | 2
  Pre-Dose 1 (Day 1) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] | 0 [0 to 33.6] | 0 [0 to 84.2]
  Post-Dose 1 Day 7 (Day 8) | 25 [5.5 to 57.2] | 58 [27.7 to 84.8] | 0 [0 to 45.9] | 0 [0 to 26.5] | 20 [2.5 to 55.6] | 17 [0.4 to 64.1] | 58 [27.7 to 84.8] | 0 [0 to 70.8]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] | 17 [2.1 to 48.4] | 0 [0 to 70.8]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 17 [2.1 to 48.4] | 17 [2.1 to 48.4] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] | 83 [51.6 to 97.9] | 0 [0 to 70.8]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 8 [0.2 to 38.5] | 17 [2.1 to 48.4] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] |  |

14. Secondary Outcome: Percentage of Participants With >= 2-fold Rise in ALS Anti-dmLT-specific IgA Titers Over Baseline Measured by ELISA
Description: Blood was collected for the IgA and IgG assay which was conducted with dmLT as the antigen. Each sample was tested per the laboratory's standard operating procedure. The percentage of participants with a >= 2-fold rise in ALS anti-dmLT-specific IgG and IgA titers over baseline was calculated for each study arm from the available results at any time post-first study vaccination.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 1 through Day 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Post-Dose 1 Day 7 (Day 8) | 75 [42.8 to 94.5] | 100 [73.5 to 100] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] | 83 [51.6 to 97.9] | 0 [0 to 70.8]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 0 [0 to 26.5] | 17 [2.1 to 48.4] | 17 [0.4 to 64.1] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] | 58 [27.7 to 84.8] | 0 [0 to 70.8]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 42 [15.2 to 72.3] | 42 [15.2 to 72.3] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 40 [12.2 to 73.8] | 17 [0.4 to 64.1] | 92 [61.5 to 99.8] | 0 [0 to 70.8]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 0 [0 to 26.5] | 0 [0 to 26.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 25 [5.5 to 57.2] | 42 [15.2 to 72.3] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 30 [6.7 to 65.2] | 17 [0.4 to 64.1] |  |

15. Secondary Outcome: Percentage of Participants With >= 2-fold Rise in ALS Anti-dmLT-specific IgG Titers Over Baseline Measured by ELISA
Description: as for outcome 14
Time Frame: Day 1 through Day 36
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Post-Dose 1 Day 7 (Day 8) | 67 [34.9 to 90.1] | 100 [73.5 to 100] | 17 [0.4 to 64.1] | 8 [0.2 to 38.5] | 40 [12.2 to 73.8] | 0 [0 to 45.9] | 100 [73.5 to 100] | 0 [0 to 70.8]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 8 [0.2 to 38.5] | 75 [42.8 to 94.5] | 17 [0.4 to 64.1] | 8 [0.2 to 38.5] | 20 [2.5 to 55.6] | 0 [0 to 45.9] | 100 [73.5 to 100] | 33 [0.8 to 90.6]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 50 [21.1 to 78.9] | 83 [51.6 to 97.9] | 0 [0 to 45.9] | 25 [5.5 to 57.2] | 60 [26.2 to 87.8] | 0 [0 to 45.9] | 100 [73.5 to 100] | 0 [0 to 70.8]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 17 [2.1 to 48.4] | 42 [15.2 to 72.3] | 0 [0 to 45.9] | 17 [2.1 to 48.4] | 10 [0.3 to 44.5] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 42 [15.2 to 72.3] | 58 [27.7 to 84.8] | 0 [0 to 45.9] | 17 [2.1 to 48.4] | 30 [6.7 to 65.2] | 17 [0.4 to 64.1] |  |

16. Secondary Outcome: Percentage of Participants With >= 4-fold Rise Over Baseline in dmLT-specific Fecal IgA Titers Measured by ELISA
Description: Stool was collected for the IgA assay which was conducted with dmLT as the antigen. Each sample was tested per the laboratory's standard operating procedure. The percentage of participants with a >= 4-fold rise over baseline in dmLT-specific fecal IgA titers was calculated for each study arm from the available results at any time post-first study vaccination.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 1 through Day 57
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Post-Dose 1 Day 7 (Day 8) | 0 [0 to 26.5] | 25 [5.5 to 57.2] | 0 [0 to 45.9] | 17 [2.1 to 48.4] | 40 [12.2 to 73.8] | 17 [0.4 to 64.1] | 8 [0.2 to 38.5] | 67 [9.4 to 99.2]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 25 [5.5 to 57.2] | 33 [9.9 to 65.1] | 17 [0.4 to 64.1] | 17 [2.1 to 48.4] | 30 [6.7 to 65.2] | 33 [4.3 to 77.7] | 0 [0 to 26.5] | 33 [0.8 to 90.6]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 8 [0.2 to 38.5] | 58 [27.7 to 84.8] | 17 [0.4 to 64.1] | 8 [0.2 to 38.5] | 20 [2.5 to 55.6] | 33 [4.3 to 77.7] | 0 [0 to 26.5] | 33 [0.8 to 90.6]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 25 [5.5 to 57.2] | 33 [9.9 to 65.1] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 30 [6.7 to 65.2] | 50 [11.8 to 88.2] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 25 [5.5 to 57.2] | 33 [9.9 to 65.1] | 17 [0.4 to 64.1] | 8 [0.2 to 38.5] | 30 [6.7 to 65.2] | 17 [0.4 to 64.1] |  |
  Post-Dose 3 Day 28 (Day 57 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 11 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 28 (Day 57 oral/sublingual) | 25 [5.5 to 57.2] | 42 [15.2 to 72.3] | 17 [0.4 to 64.1] | 27 [6.0 to 61.0] | 20 [2.5 to 55.6] | 33 [4.3 to 77.7] |  |

17. Secondary Outcome: Percentage of Participants With >= 4-fold Rise Over Baseline in dmLT-specific Salivary IgA Titers Measured by ELISA
Description: Saliva was collected for the IgA assay which was conducted with dmLT as the antigen. Each sample was tested per the laboratory's standard operating procedure. The percentage of participants with a >= 4-fold rise over baseline in dmLT-specific salivary IgA titers was calculated for each study arm from the available results at any time post-first study vaccination.
  Study halted on Day 43 due to COVID-19 pandemic and the intradermal group did not receive the final dose.
Time Frame: Day 1 through Day 57
Population: as for outcome 12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 12 | 3
percentage of participants
  Post-Dose 1 Day 7 (Day 8) | 0 [0 to 26.5] | 8 [0.2 to 38.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 33 [0.8 to 90.6]
  Pre-Dose 2 (Day 15 oral/sublingual, Day 22 intradermal) | 8 [0.2 to 38.5] | 17 [2.1 to 48.4] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 30.8] | 0 [0 to 45.9] | 0 [0 to 26.5] | 0 [0 to 70.8]
  Post-Dose 2 Day 7 (Day 22 oral/sublingual, Day 29 intradermal) | 0 [0 to 26.5] | 8 [0.2 to 38.5] | 0 [0 to 45.9] | 0 [0 to 26.5] | 10 [0.3 to 44.5] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 33 [0.8 to 90.6]
  Pre-Dose 3 (Day 29 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Pre-Dose 3 (Day 29 oral/sublingual) | 8 [0.2 to 38.5] | 17 [2.1 to 48.4] | 0 [0 to 45.9] | 8 [0.2 to 38.5] | 0 [0 to 30.8] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 7 (Day 36 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 7 (Day 36 oral/sublingual) | 0 [0 to 26.5] | 8 [0.2 to 38.5] | 0 [0 to 45.9] | 17 [2.1 to 48.4] | 0 [0 to 30.8] | 0 [0 to 45.9] |  |
  Post-Dose 3 Day 28 (Day 57 oral/sublingual): number analyzed (Participants) | 12 | 12 | 6 | 12 | 10 | 6 | 0 | 0
  Post-Dose 3 Day 28 (Day 57 oral/sublingual) | 8 [0.2 to 38.5] | 17 [2.1 to 48.4] | 0 [0 to 45.9] | 9 [0.2 to 41.3] | 0 [0 to 30.8] | 0 [0 to 45.9] |  |

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected for 7 days after each vaccine administration. Unsolicited AEs were collected from the time of each study vaccination through 28 days after the last vaccination. Serious adverse events (SAEs) were collected from the time of the first study vaccination through 6 months after the last study vaccination.
Description: Solicited AEs include local and systemic. Systemic reactions include feverishness, fatigue, myalgia, headache, diarrhea, nausea, vomiting or abdominal discomfort and temperature. Local reactions for oral and sublingual include irritation of oral cavity or tongue, diarrhea, nausea, vomiting, and abdominal discomfort. Local reactions for intradermal include injection site pain, redness, swelling, bruising, itching, hypo/hyper pigmentation and induration, and vesicles or hardened mass.
Arm/Group | Oral 5 µg dmLT | Oral 25 µg of dmLT | Oral Placebo | Sublingual 5 µg of dmLT | Sublingual 25 µg of dmLT | Sublingual Placebo | Intradermal 0.3 µg of dmLT | Intradermal Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/6 | 0/12 | 0/12 | 0/6 | 0/12 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/6 | 0/12 | 0/12 | 0/6 | 0/12 | 0/3
Other Adverse Events (participants affected / at risk) | 1/12 | 0/12 | 1/6 | 0/12 | 4/12 | 0/6 | 0/12 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral 5 µg dmLT (N=12) | Oral 25 µg of dmLT (N=12) | Oral Placebo (N=6) | Sublingual 5 µg of dmLT (N=12) | Sublingual 25 µg of dmLT (N=12) | Sublingual Placebo (N=6) | Intradermal 0.3 µg of dmLT (N=12) | Intradermal Placebo (N=3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropihl count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03548064/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT03548064/SAP_002.pdf
  • Informed Consent Form (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT03548064/ICF_001.pdf